CLINICAL TRIAL: NCT06307418
Title: The Effects of Internet-based Support (Carer eSupport) on Preparedness for Caregiving in Informal Caregivers of Patients With Head and Neck Cancer Compared to Standard Care Support - a Study Protocol for a Randomized Controlled Trial
Brief Title: Internet-based Support for Informal Caregivers of Patients With Head and Neck Cancer - Carer eSupport
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Cancer Society (Other); Umeå University (Other); Region Örebro County (Other); Sahlgrenska University Hospital (Other); University Hospital, Umeå (Other); Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Birgitta Johansson, Senior lecturer, Associate professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Carer eSupport RCT
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer
Keywords: Informal caregivers; Internet-based support; Preparedness for caregiving; Caregiver burden; Quality of life
MeSH Terms: conditions — Head and Neck Neoplasms; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Informal caregivers of patients with Head and neck cancer will be randomized to internet-based support or to support as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based support (Carer eSupport) (Experimental): The internet-based support is developed in collaboration with clinical expertise within head and neck cancer care and an expert group of informal caregivers to patients with head and neck cancer. The support comprise text, lectures, films, discussion forum and real-time video meetings with clinical experts. The support will last for 18 weeks.
  Interventions: Other: Carer eSupport
- Support as usual (No Intervention): Support as usual comprise a possibility for informal caregivers to contact a specified nurse with expertise in head and neck , at the head and neck or oncology clinic, to ask for support. Healthcare counsellors at the clinics is also available for ICs on request. Group support providing emotional and social support for ICs to patients with various cancer diagnoses may also be arranged at the clinics occasionally. Also, the Swedish healthcare is always responsible for recognizing the need for support for children (< 18 years) of patients with cancer.

INTERVENTIONS:
Other: Carer eSupport — Internet-based support
  Arms: Internet-based support (Carer eSupport)

SUMMARY:
The aim of this randomized controlled trial is to investigate the effects of internet-based support (Carer eSupport) on preparedness for caregiving in informal caregivers of patients with head and neck cancer. The main question[s] it aims to answer are:

* What are the effects of internet-based support on informal caregivers preparedness for caregiving?
* What are the effects of internet-based support on informal caregivers burden and wellbeing?

Informal caregivers who are randomized to Carer eSupport will have access to Carer eSupport for 18 weeks and they will be asked to complete questionnaires (outcome measures) at:

* baseline (before randomization)
* 18 weeks (post-intervention) and at
* 3 months after the intervention is completed (long term follow-up).

Informal caregivers in the intervention group will be compared to informal caregivers who receive standard care support regarding preparedness for caregiving, caregiver burden and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers who have been identified as an informal caregiver by a patient who have consented to that the informal caregivers is approached.
* Informal caregivers of patients with head and neck cancer who are about to start radiotherapy or have undergone at most five radiotherapy treatment session. Radiotherapy may be combined with surgery and/or medical oncological treatment.

Exclusion Criteria:

* Informal caregivers who do not understand and read Swedish or suffer from cognitive impairment, and informal caregivers with who need support or treatment that cannot be provided by Carer eSupport.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
The self-reported questionnaire Preparedness for caregiving scale | Baseline, 18 weeks after randomization (post-intervention) and 3 months after post-intervention.
  A self-reported questionnaire consisting of eight items, responded to on a 5-grade scale (0 not at all prepared - 4 very well prepared) concerning informal caregivers' (ICs) self-reported preparedness to take care of the patient's needs, find out about and set up services, get support from the health care system and manage the stress related to being an informal caregiver. The scores are summed to a scale ranging from 0-32, with a higher score reflecting better preparedness.

SECONDARY OUTCOMES:
The self-reported questionnaire Caregiver Burden Scale | Baseline, 18 weeks after randomization (post-intervention) and 3 months after post-intervention.
  A self-reported questionnaire consisting of 22 items responded to on a 4-grade scale (1 Not at all - 4 Often), a higher score indicates a more significant burden. The 22 items may be divided into the factors of General strain, Disappointment, Emotional involvement, Environment, and Isolation, and the mean of all items indicates the total burden.
The self-reported questionnaire Depression Anxiety Stress Scale-21 (DASS21) | Baseline, 18 weeks after randomization (post-intervention) and 3 months after post-intervention.
  A self-reported questionnaire consisting of 21 items constituting three subscales, with seven item each, measuring depression, anxiety, and stress. Each item is scored on a 4-grade scale, with higher scores indicating more symptoms.
The self-reported health-related quality of life questionnaire RAND-36 | Baseline, 18 weeks after randomization (post-intervention) and 3 months after post-intervention.
  A self-reported health-related quality of life questionnaire consisting of 36 items measuring physical functioning (10 items), role limitations due to physical (4 items) and emotional (3 items) health problems, social functioning (2 items), emotional well-being (5 items), energy/fatigue (4 items), pain (2 items), and general health perceptions (5 items) and perceived change in health (1 item). All scales are scored so that that the lowest and highest possible scores are set at 0 and 100, respectively. Higher scores indicate a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Tiblom Ehrsson, Assoc prof, Principal Investigator — Uppsala University
Locations (4):
- Sweden (4):
  - Örebro University Hospital, Örebro, Blekinge Län
  - Uppsala university hospital, Uppsala, Uppsala County
  - Norrland University Hospital, Umeå, Västerbotten County
  - Sahlgrenska university hospital, Gothenburg, Västra Götaland County

REFERENCES:
- [Derived] Johansson B, Cajander A, Ahmad A, Ohlsson-Nevo E, Fransson P, Granstrom B, von Essen L, Langegard U, Pettersson M, Henriksson A, Ehrsson YT. The effect of internet-administered support (carer eSupport) on preparedness for caregiving in informal caregivers of patients with head and neck cancer compared with support as usual: a study protocol for a randomized controlled trial. BMC Cancer. 2024 Apr 18;24(1):494. doi: 10.1186/s12885-024-12273-y. PMID 38637744